CLINICAL TRIAL: NCT02171611
Title: Relative Bioavailability of Dabigatran After Administration of Different Application Forms of a Single Oral Dose of 150 mg Dabigatran Etexilate (Capsule, Powder for Reconstitution Into Solution, Pellets on Food) in Healthy Male and Female Volunteers (an Open-label, Randomised, Three-way Crossover, Clinical Phase I Study)
Brief Title: Bioavailability of Different Applications of Dabigatran in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.87
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran

ARMS (3):
- Dabigatran etexilate pellets (Experimental)
  Interventions: Drug: Dabigatran etexilate pellets
- Dabigatran etexilate powder (Experimental)
  Interventions: Drug: Dabigatran etexilate powder
- Dabigatran etexilate capsule (Active Comparator)
  Interventions: Drug: Dabigatran etexilate capsule

INTERVENTIONS:
Drug: Dabigatran etexilate pellets
  Arms: Dabigatran etexilate pellets
Drug: Dabigatran etexilate powder
  Arms: Dabigatran etexilate powder
Drug: Dabigatran etexilate capsule
  Arms: Dabigatran etexilate capsule

SUMMARY:
To determine the relative bioavailability of 150 mg of dabigatran etexilate as pellets on food and of 150 mg of dabigatran etexilate as powder resolved in reconstitution solution, both with 150 mg of dabigatran etexilate as capsule in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
* Age ≥18 and age ≤50 years
* BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which could reasonably influence the results of the trial (especially unspecific inducing agents like St. John´s wort (Hypericum perforatum) or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that was of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g. repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for Torsade de Pointes (e.g. heart failure, hypokalemia, family history of Long QT Syndrome)
* For female subjects:

  * Positive pregnancy test, pregnancy or planning to become pregnant during the study or within 1 month after study completion
  * No adequate contraception during the study and until 1 month after study completion, i.e. not any of the following: implants, injectables, combined oral contraceptives, intrauterine device (IUD), sexual abstinence for at least 1 month prior to enrolment, vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilisation (including hysterectomy). Females, who did not have a vasectomised partner, were not sexually abstinent or surgically sterile were to be asked to use an additional barrier method (e.g. condom, diaphragm with spermicide)
  * Lactation
* Intake of medication, which influences the blood clotting, i.e. acetylsalicylic acid, oral vitamin K antagonists etc.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- A/B/C: Subjects were treated after an overnight fast of at least 10 hours with single oral dose, started in Period 1 with Dabigatran etexilate 150 mg capsule: Reference (A) with about 240 mL of water and in Period 2 with Dabigatran etexilate 150 mg pellets: Test 1 (B) by sprinkling the pellets on a teaspoon of food and administered immediately to the subject, followed in period 3 with Dabigatran etexilate 150 mg powder: Test 2 (C) resolved in 24 mL reconstitution solution.
  Treatments were separated by washout period of at least 7 days after drug administration.
- A/C/B: Subjects were treated after an overnight fast of at least 10 hours with single oral dose, started in Period 1 with Dabigatran etexilate 150 mg capsule: Reference (A) with about 240 mL of water and in period 2 with Dabigatran etexilate 150 mg powder: Test 2 (C) resolved in 24 mL reconstitution solution, followed in Period 3 with Dabigatran etexilate 150 mg pellets: Test 1 (B) by sprinkling the pellets on a teaspoon of food and administered immediately to the subject.
  Treatments were separated by washout period of at least 7 days after drug administration.
- B/A/C: Subjects were treated after an overnight fast of at least 10 hours with single oral dose, started in Period 1 with Dabigatran etexilate 150 mg pellets: Test 1 (B) by sprinkling the pellets on a teaspoon of food and administered immediately to the subject and in period 2 with Dabigatran etexilate 150 mg capsule: Reference (A) with about 240 mL of water, followed in Period 3 with Dabigatran etexilate 150 mg powder: Test 2 (C) resolved in 24 mL reconstitution solution.
  Treatments were separated by washout period of at least 7 days after drug administration.
- B/C/A: Subjects were treated after an overnight fast of at least 10 hours with single oral dose, started in Period 1 with Dabigatran etexilate 150 mg pellets: Test 1 (B) by sprinkling the pellets on a teaspoon of food and administered immediately to the subject and in period 2 with Dabigatran etexilate 150 mg powder: Test 2 (C) resolved in 24 mL reconstitution solution, followed in period 3 with Dabigatran etexilate 150 mg capsule: Reference (A) with about 240 mL of water.
  Treatments were separated by washout period of at least 7 days after drug administration.
- C/A/B: Subjects were treated after an overnight fast of at least 10 hours with single oral dose, started in Period 1 with Dabigatran etexilate 150 mg powder: Test 2 (C) resolved in 24 mL reconstitution solution and in period 2 with Dabigatran etexilate 150 mg capsule: Reference (A) with about 240 mL of water, followed in Period 3 with Dabigatran etexilate 150 mg pellets: Test 1 (B) by sprinkling the pellets on a teaspoon of food and administered immediately to the subject. Treatments were separated by washout period of at least 7 days after drug administration.
- C/B/A: Subjects were treated after an overnight fast of at least 10 hours with single oral dose, started in Period 1 with Dabigatran etexilate 150 mg powder: Test 2 (C) resolved in 24 mL reconstitution solution and in period 2 with Dabigatran etexilate 150 mg pellets: Test 1 (B) by sprinkling the pellets on a teaspoon of food and administered immediately to the subject, followed in Period 3 with Dabigatran etexilate 150 mg capsule: Reference (A) with about 240 mL of water.
  Treatments were separated by washout period of at least 7 days after drug administration.
Period: Overall Study
Arm/Group | A/B/C | A/C/B | B/A/C | B/C/A | C/A/B | C/B/A
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This subject set included all subjects who were dispensed trial medication and were documented to have taken at least one dose of investigational treatment. This set was used for safety analysis.
Groups:
- Overall: This study is open-label, single dose, randomised, three-way crossover design having 3 treatment periods ie., Dabigatran etexilate 150 mg formulation capsule: Reference (A), Dabigatran etexilate 150 mg formulation pellets: Test 1 (B) and Dabigatran etexilate 150 mg formulation powder: Test 2 (C)
Arm/Group | Overall
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: AUC0-inf for Total Dabigatran
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf) for total dabigatran.
Time Frame: -0:30 hour(h) before drug administration and 0:30h, 1:00h, 1:30h, 2:00h, 2:30h, 3:00h, 3:30h, 4:00h, 6:00h, 8:00h, 12:00h, 24:00h, 36:00h and 48:00h after drug administration.
Population: PK-Per protocol set (PK-PPS): This subject set included all subjects in the treated set who provided at least one observation for at least one primary (PK) endpoint without important protocol violations with respect to the evaluation of relative bioavailability and who did not vomit at or before 2 times the median tmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng(nanogram)*h(hour)/mL(milliliter)
Groups:
- Dabigatran Etexilate 150 mg Capsule: Reference (A): Subjects were treated with single oral dose of Dabigatran etexilate 150 mg formulation capsule: Reference (A) after an overnight fast of at least 10 hours with about 240 milliliter (mL) of water.
- Dabigatran Etexilate 150 mg Pellets: Test 1 (B): Subjects were treated with single oral dose of Dabigatran etexilate 150 mg formulation pellets: Test 1 (B) after an overnight fast of at least 10 hours. Pellets were sprinkled on a teaspoon of food and administered immediately to the subject.
- Dabigatran Etexilate 150 mg Powder: Test 2 (C): Subjects were treated with single oral dose of Dabigatran etexilate 150 mg formulation powder: Test 2 (C) resolved in 24 mL reconstitution solution after an overnight fast of at least 10 hours.
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
ng(nanogram)*h(hour)/mL(milliliter) | 599 (93.3) | 1050 (33.8) | 928 (32.8)
Statistical Analysis 1: Comparison: Dabigatran Etexilate 150 mg Capsule: Reference (A) vs Dabigatran Etexilate 150 mg Pellets: Test 1 (B); An Analysis of variance (ANOVA) model was used on the logarithmic scale in order to compare the Test treatment vs. the Reference treatment. This model included effects for 'sequence', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Test type: Superiority or Other; Ratio of adjusted geometric means = 175.14, 90% CI 2-sided [141.904 to 216.149], Standard Error of Mean 50.7 — Relative bioavailability was estimated by the ratio of the gMeans of Dabigatran etexilate 150 mg (T1) divided by Dabigatran etexilate 150 mg (R). Standard Error of the mean is actually the intra individual coefficient variation (gCV)
Statistical Analysis 2: Comparison: Dabigatran Etexilate 150 mg Capsule: Reference (A) vs Dabigatran Etexilate 150 mg Powder: Test 2 (C); An Analysis of variance (ANOVA) model was used on the logarithmic scale in order to compare the Test treatment (T2) vs. the Reference treatment (R). This model included effects for 'sequence', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Test type: Superiority or Other; Ratio of adjusted geometric means = 154.84, 90% CI 2-sided [127.425 to 188.161], Standard Error of Mean 46.6 — Relative bioavailability was estimated by the ratio of the geometric means (gMeans) of Dabigatran etexilate 150 mg (T2) divided by Dabigatran etexilate 150 mg (R). Standard Error of the mean is actually the intra individual gCV

2. Primary Outcome: AUC0-inf for Free Dabigatran
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf) for free dabigatran.
Time Frame: as for outcome 1
Population: pharmacokinetic per-protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
ng*h/mL | 464 (97.3) | 815 (40) | 734 (38.2)
Statistical Analysis 1: Comparison: Dabigatran Etexilate 150 mg Capsule: Reference (A) vs Dabigatran Etexilate 150 mg Pellets: Test 1 (B); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio of adjusted geometric means in % = 175.4, 90% CI 2-sided [141.924 to 216.772], Standard Error of Mean 51.1 — Relative bioavailability was estimated by the ratio of the gMean of Dabigatran etexilate 150 mg (T1) divided by Dabigatran etexilate 150 mg (R). Standard Error of the mean is actually the intra individual gCV
Statistical Analysis 2: Comparison: Dabigatran Etexilate 150 mg Capsule: Reference (A) vs Dabigatran Etexilate 150 mg Powder: Test 2 (C); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio of adjusted geometric means in % = 158.12, 90% CI 2-sided [130.052 to 192.255], Standard Error of Mean 46.7 — Relative bioavailability was estimated by the ratio of the gMean of Dabigatran etexilate 150 mg (T2) divided by Dabigatran etexilate 150 mg (R). Standard Error of the mean is actually the intra individual gCV

3. Primary Outcome: Cmax for Total Dabigatran
Description: Maximum measured concentration of the analyte in plasma (Cmax) for total dabigatran.
Time Frame: as for outcome 1
Population: pharmacokinetic per-protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
ng/mL | 74.6 (110) | 139 (37.8) | 124 (37)
Statistical Analysis 1: Comparison: Dabigatran Etexilate 150 mg Capsule: Reference (A) vs Dabigatran Etexilate 150 mg Pellets: Test 1 (B); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio of adjusted geometric means = 186.94, 90% CI 2-sided [147.659 to 236.665], Standard Error of Mean 57.7 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Dabigatran Etexilate 150 mg Capsule: Reference (A) vs Dabigatran Etexilate 150 mg Powder: Test 2 (C); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio of adjusted geometric means in % = 166.59, 90% CI 2-sided [133.221 to 208.326], Standard Error of Mean 54.3 — [estimate comment as in outcome 2, analysis 2]

4. Primary Outcome: Cmax for Free Dabigatran
Description: Maximum measured concentration of the analyte in plasma (Cmax) for free dabigatran
Time Frame: as for outcome 1
Population: pharmacokinetic per-protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
ng/mL | 61.5 (110) | 112 (40.4) | 103 (40.7)
Statistical Analysis 1: Comparison: Dabigatran Etexilate 150 mg Capsule: Reference (A) vs Dabigatran Etexilate 150 mg Pellets: Test 1 (B); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio of adjusted geometric means in % = 181.6, 90% CI 2-sided [145.428 to 226.776], Standard Error of Mean 53.9 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Dabigatran Etexilate 150 mg Capsule: Reference (A) vs Dabigatran Etexilate 150 mg Powder: Test 2 (C); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio of adjusted geometric means in % = 166.83, 90% CI 2-sided [134.25 to 207.328], Standard Error of Mean 52.6 — Relative bioavailability was estimated by the ratio of the gMean of Dabigatran etexilate 150 mg (T2) divided by Dabigatran etexilate 150 mg (R). Standard Error of the mean is actually the intra individual geometric coefficient variation (gCV)

5. Secondary Outcome: AUC0-tz for Total Dabigatran
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz) for total dabigatran.
Time Frame: as for outcome 1
Population: pharmacokinetic per-protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
ng*h/mL | 565 (106) | 1030 (34.2) | 908 (33.5)
Statistical Analysis 1: Comparison: Dabigatran Etexilate 150 mg Capsule: Reference (A) vs Dabigatran Etexilate 150 mg Pellets: Test 1 (B); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio of adjusted geometric means in % = 182.17, 90% CI 2-sided [144.727 to 229.297], Standard Error of Mean 56.1 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Dabigatran Etexilate 150 mg Capsule: Reference (A) vs Dabigatran Etexilate 150 mg Powder: Test 2 (C); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio of adjusted geometric means in % = 160.74, 90% CI 2-sided [129.633 to 199.306], Standard Error of Mean 52 — [estimate comment as in outcome 2, analysis 2]

6. Secondary Outcome: AUC0-tz for Free Dabigatran
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz) for free dabigatran.
Time Frame: as for outcome 1
Population: pharmacokinetic per-protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
ng*h/mL | 436 (110) | 794 (41.3) | 715 (39.5)
Statistical Analysis 1: Comparison: Dabigatran Etexilate 150 mg Capsule: Reference (A) vs Dabigatran Etexilate 150 mg Pellets: Test 1 (B); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio of adjusted geometric means in % = 182.25, 90% CI 2-sided [144.993 to 229.075], Standard Error of Mean 55.7 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Dabigatran Etexilate 150 mg Capsule: Reference (A) vs Dabigatran Etexilate 150 mg Powder: Test 2 (C); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio of adjusted geometric means in % = 164.01, 90% CI 2-sided [132.421 to 203.14], Standard Error of Mean 51.7 — [estimate comment as in outcome 2, analysis 2]

7. Secondary Outcome: Tmax for Total Dabigatran
Description: Time from dosing to the maximum concentration of the analyte in plasma (tmax) for total dabigatran
Time Frame: as for outcome 1
Population: pharmacokinetic per-protocol set
Measure: Median (Full Range); unit: hour
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
hour | 2.0 [1.5 to 6.0] | 1.5 [1.0 to 3.0] | 1.5 [1.0 to 2.5]

8. Secondary Outcome: Tmax for Free Dabigatran
Description: Time from dosing to the maximum concentration of the analyte in plasma (tmax) for free dabigatran
Time Frame: as for outcome 1
Population: pharmacokinetic per-protocol set
Measure: Median (Full Range); unit: hour
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
hour | 2.0 [1.5 to 6.0] | 1.51 [1.0 to 3.0] | 1.5 [1.0 to 2.0]

9. Secondary Outcome: λz for Total Dabigatran
Description: Terminal rate constant in plasma (λz) for total dabigatran.
Time Frame: as for outcome 1
Population: pharmacokinetic per-protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
1/hour | 0.079 (13.5) | 0.074 (14.5) | 0.0756 (16.4)

10. Secondary Outcome: λz for Free Dabigatran
Time Frame: as for outcome 1
Population: pharmacokinetic per-protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
1/hour | 0.091 (16) | 0.0811 (18.6) | 0.0893 (15.7)

11. Secondary Outcome: t1/2 for Total Dabigatran
Description: Terminal half-life of the analyte in plasma (t1/2) for total dabigatran
Time Frame: as for outcome 1
Population: pharmacokinetic per-protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
hour | 8.77 (13.5) | 9.37 (14.5) | 9.16 (16.4)

12. Secondary Outcome: t1/2 for Free Dabigatran
Description: Terminal half-life of the analyte in plasma (t1/2) for free dabigatran.
Time Frame: as for outcome 1
Population: pharmacokinetic per-protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
hour | 7.62 (16) | 8.54 (18.6) | 7.76 (15.7)

13. Secondary Outcome: MRTpo for Total Dabigatran
Description: Mean residence time of the analyte in the body after po administration (MRTpo) for total dabigatran.
Time Frame: as for outcome 1
Population: pharmacokinetic per-protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
hour | 10.8 (12) | 10.1 (11.4) | 10 (12.2)

14. Secondary Outcome: MRTpo for Free Dabigatran
Description: Mean residence time of the analyte in the body after po administration (MRTpo) for free dabigatran.
Time Frame: as for outcome 1
Population: pharmacokinetic per-protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
hour | 9.9 (14.0) | 9.58 (14.1) | 9.15 (12.2)

15. Secondary Outcome: CL/F for Total Dabigatran
Description: Apparent clearance of the analyte in plasma following extravascular administration (CL/F) for total dabigatran.
Time Frame: as for outcome 1
Population: pharmacokinetic per-protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL (milliliter)/min (minute)
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
mL (milliliter)/min (minute) | 3130 (93.3) | 1790 (33.8) | 2020 (32.8)

16. Secondary Outcome: CL/F for Free Dabigatran
Description: Apparent clearance of the analyte in plasma following extravascular administration (CL/F) for free dabigatran.
Time Frame: as for outcome 1
Population: pharmacokinetic per-protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL (milliliter)/min (minute)
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
mL (milliliter)/min (minute) | 4040 (97.3) | 2310 (40) | 2560 (38.2)

17. Secondary Outcome: Vz/F for Total Dabigatran
Description: Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F) for total dabigatran.
Time Frame: as for outcome 1
Population: pharmacokinetic per-protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
Liter | 2380 (92.8) | 1450 (35) | 1610 (35.9)

18. Secondary Outcome: Vz/F for Free Dabigatran
Description: Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F) for free dabigatran.
Time Frame: as for outcome 1
Population: pharmacokinetic per-protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
Liter | 2670 (91) | 1700 (41.4) | 1720 (37.6)

19. Secondary Outcome: Percentage of Participants With Findings in Physical Examination, Vital Signs , Pulse Rate (PR)), 12-lead ECG, Clinical Laboratory Tests.
Description: Percentage of participants with findings in Physical examination, Vital signs (blood pressure (BP), pulse rate (PR)), 12-lead ECG (electrocardiogram), Clinical laboratory tests (haematology, clinical chemistry and urinalysis). Relevant findings or worsening of baseline conditions were reported as Adverse events.
  There were no clinically relevant finding reported for Physical examination, Vital signs (blood pressure, pulse rate), 12-lead ECG and Clinical laboratory tests.
Time Frame: From first drug administration until 7 days after the last drug administration of Dabigatran, ie., up to 10 days.
Population: Treated Set
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
Percentage of participants | 0.0 | 0.0 | 0.0

20. Secondary Outcome: Percentage of Participants With Drug-related Adverse Events
Description: Percentage of participants with investigator defined drug-releated Adverse events.
Time Frame: From first drug administration until 7 days after the last drug administration of Dabigatran, ie., up to 10 days.
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
Percentage of participants | 6.7 | 23.3 | 26.7

21. Secondary Outcome: Assessment of Tolerability by Investigator.
Description: Tolerability will be assessed by the investigator according to the categories good, satisfactory, not satisfactory and bad.
Time Frame: From first drug administration until 7 days after the last drug administration of Dabigatran, ie., up to 10 days.
Population: Treated Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Number analyzed (Participants) | 30 | 30 | 30
Percentage of Participants
  Good | 100.0 | 100.0 | 100.0
  Satisfactory | 0.0 | 0.0 | 0.0
  Not satisfactory | 0.0 | 0.0 | 0.0
  Bad | 0.0 | 0.0 | 0.0
  Not assessable | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: From first drug administration until 7 days after the last drug administration of Dabigatran, ie., up to 10 days.
Arm/Group | Dabigatran Etexilate 150 mg Capsule: Reference (A) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) | Dabigatran Etexilate 150 mg Powder: Test 2 (C)
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 2/30 | 7/30 | 8/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate 150 mg Capsule: Reference (A) (N=30) | Dabigatran Etexilate 150 mg Pellets: Test 1 (B) (N=30) | Dabigatran Etexilate 150 mg Powder: Test 2 (C) (N=30)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 2 | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.